CLINICAL TRIAL: NCT04115982
Title: Vitamin D3 in Sensory Recovery After Digital NERVe Suture: a Randomized Controlled Trial.
Brief Title: Vitamin D3 in Sensory Recovery After Digital NERVe Suture (D3NERV).
Acronym: D3NERV
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-237; 2018-001526-26 (EudraCT Number)
Record Dates: First submitted 2019-08-19; First posted 2019-10-04 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-07

CONDITIONS: Digital Nerve Injury
Keywords: digital nerve injury; neuroma; cholecalciferol
MeSH Terms: conditions — Neuroma | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cholecalciferol (Experimental): Cholecalciferol (Vitamin D3) 100 000 IU/2 mL
  Interventions: Drug: Cholecalciferol
- Placebo (Placebo Comparator): Placebo of Cholecalciferol (Vitamine D3) 100 000 IU/2 mL
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Cholecalciferol — One vial every 15 days during 2 months
  Arms: Cholecalciferol
Drug: Placebos — One vial every 15 days during 2 months
  Arms: Placebo

SUMMARY:
Digital nerve injuries are frequent in a FESUM center (Federation Européenne des Services d'Urgences Mains), and they need to be repaired in order to reduce the risk of hypoesthesia and to prevent painful neuroma. Several animal studies have shown that Cholecalciferol improves axonal nerve regeneration and myelination. No study has ever been done on human subjects to evaluate the nerve regeneration after Cholecalciferol supplementation.

Our hypothesis is that Cholecalciferol supplementation could improve axonal nerve regeneration and myelination after traumatic digital nerve injuries treated by microsurgical sutures and reduce the risk of hypoesthesia and neuroma.

ELIGIBILITY:
Inclusion Criteria:

* Affiliated to social security scheme,
* Wound of the palmar hand with isolated digital nerve section, requiring digital nerve microsurgical suture in the operating room by a senior surgeon,
* Signing a free and informed consent and well-informed of the study and procedure.

Exclusion Criteria:

* Ischemia,
* Multiple lesion of the same nerve,
* Pregnant or nursing women,
* Contraindication of Cholecalciferol : known hypersensitivity, any history of hypercalcemia, hypercalciuria or renal lithiasis,
* Cholecalciferol supplementation in the past 6 months,
* Lesion of the same controlateral finger,
* History of nerve lesion or hypoesthesia on the same finger,
* History of previous neurological disorders with upper limb sensitivity disorder,
* Impossibility to undergo the medical follow-up because of geographical, social or psychological reason,
* Participation in another clinical trial that does not allow simultaneous participation in several clinical trials,
* Orlistat® Treatment,
* History of celiac disease.

Ages: 18 Years to 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Weber test (Month 6) | Month 6
  2 point discrimination test of Weber on the side of the fingertip concerned by the wound, comparing to the controlateral arm, after 6 months.

SECONDARY OUTCOMES:
Weber test (Month 12) | Month 12
  2 point discrimination test of Weber on the side of the fingertip concerned by the wound, comparing to the controlateral arm, after 12 months.
Resting pain on the operated finger | Month 2, Month 6, Month 12
  VAS (Visual Analogic Scale)
Neuropathic pain on the operated finger | Month 2, Month 6, Month 12
  DN 4 (Neuropathic pain)
Global functional outcome measure | Month 2, Month 6, Month 12
  Quick DASH
Cold Intolerance | Month 2, Month 6, Month 12
  CSS (Cold Sensitivity Severity Scale)
Cold Intolerance at work | Month 2, Month 6, Month 12
  PWES (Potential Work Exposure Scale)
Quality-of-life measure | Month 2, Month 6, Month 12
  SF-36 (Study Short form 36)
Return-to-work time frames | Month 2
  Time before returning to work
Vitamin D blood level | at inclusion, Month 2
Adverse event and complication | Trough study completion
  Existence of neuroma, existence of medical complication, existence of overdosage of Cholecalciferol and every other adverse event

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Caen University Hospital, Caen
  - Rouen University Hospital, Rouen
  - Institut de la main Nantes Atlantique, Saint-Herblain

REFERENCES:
- [Background] al-Ghazal SK, McKiernan M, Khan K, McCann J. Results of clinical assessment after primary digital nerve repair. J Hand Surg Br. 1994 Apr;19(2):255-7. doi: 10.1016/0266-7681(94)90180-5. PMID 8014564
- [Background] Alligand-Perrin P, Rabarin F, Jeudy J, Cesari B, Saint-Cast Y, Fouque PA, Raimbeau G. Vein conduit associated with microsurgical suture for complete collateral digital nerve severance. Orthop Traumatol Surg Res. 2011 Jun;97(4 Suppl):S16-20. doi: 10.1016/j.otsr.2011.03.012. Epub 2011 Apr 30. PMID 21531189
- [Background] Arnaout A, Fontaine C, Chantelot C. Sensory recovery after primary repair of palmar digital nerves using a Revolnerv((R)) collagen conduit: a prospective series of 27 cases. Chir Main. 2014 Sep;33(4):279-85. doi: 10.1016/j.main.2014.05.002. Epub 2014 Jun 18. PMID 25169199
- [Background] Barrueto F Jr, Wang-Flores HH, Howland MA, Hoffman RS, Nelson LS. Acute vitamin D intoxication in a child. Pediatrics. 2005 Sep;116(3):e453-6. doi: 10.1542/peds.2004-2580. PMID 16140692
- [Background] Battiston B, Geuna S, Ferrero M, Tos P. Nerve repair by means of tubulization: literature review and personal clinical experience comparing biological and synthetic conduits for sensory nerve repair. Microsurgery. 2005;25(4):258-67. doi: 10.1002/micr.20127. PMID 15934044
- [Background] Bertleff MJ, Meek MF, Nicolai JP. A prospective clinical evaluation of biodegradable neurolac nerve guides for sensory nerve repair in the hand. J Hand Surg Am. 2005 May;30(3):513-8. doi: 10.1016/j.jhsa.2004.12.009. PMID 15925161
- [Background] Chabas JF, Stephan D, Marqueste T, Garcia S, Lavaut MN, Nguyen C, Legre R, Khrestchatisky M, Decherchi P, Feron F. Cholecalciferol (vitamin D(3)) improves myelination and recovery after nerve injury. PLoS One. 2013 May 31;8(5):e65034. doi: 10.1371/journal.pone.0065034. Print 2013. PMID 23741446
- [Background] Heaney RP, Davies KM, Chen TC, Holick MF, Barger-Lux MJ. Human serum 25-hydroxycholecalciferol response to extended oral dosing with cholecalciferol. Am J Clin Nutr. 2003 Jan;77(1):204-10. doi: 10.1093/ajcn/77.1.204. PMID 12499343
- [Background] Neubrech F, Heider S, Otte M, Hirche C, Kneser U, Kremer T. [Nerve Tubes for the Repair of Traumatic Sensory Nerve Lesions of the Hand: Review and Planning Study for a Randomised Controlled Multicentre Trial]. Handchir Mikrochir Plast Chir. 2016 Jun;48(3):148-54. doi: 10.1055/s-0042-104505. Epub 2016 Jun 16. German. PMID 27311073
- [Background] Finnell JT, Knopp R, Johnson P, Holland PC, Schubert W. A calibrated paper clip is a reliable measure of two-point discrimination. Acad Emerg Med. 2004 Jun;11(6):710-4. PMID 15175216
- [Background] Gueye Y, Marqueste T, Maurel F, Khrestchatisky M, Decherchi P, Feron F. Cholecalciferol (vitamin D(3)) improves functional recovery when delivered during the acute phase after a spinal cord trauma. J Steroid Biochem Mol Biol. 2015 Nov;154:23-31. doi: 10.1016/j.jsbmb.2015.06.007. Epub 2015 Jul 6. PMID 26159913
- [Background] Barger-Lux MJ, Heaney RP. Effects of above average summer sun exposure on serum 25-hydroxyvitamin D and calcium absorption. J Clin Endocrinol Metab. 2002 Nov;87(11):4952-6. doi: 10.1210/jc.2002-020636. PMID 12414856
- [Background] Lundborg G, Rosen B. The two-point discrimination test--time for a re-appraisal? J Hand Surg Br. 2004 Oct;29(5):418-22. doi: 10.1016/j.jhsb.2004.02.008. PMID 15336741
- [Background] Fakin RM, Calcagni M, Klein HJ, Giovanoli P. Long-term clinical outcome after epineural coaptation of digital nerves. J Hand Surg Eur Vol. 2016 Feb;41(2):148-54. doi: 10.1177/1753193415578986. Epub 2015 Mar 31. PMID 25827143
- [Background] Manoli T, Schiefer JL, Schulz L, Fuchsberger T, Schaller HE. Influence of immobilization and sensory re-education on the sensory recovery after reconstruction of digital nerves with direct suture or muscle-in-vein conduits. Neural Regen Res. 2016 Feb;11(2):338-44. doi: 10.4103/1673-5374.169638. PMID 27073390
- [Background] Montava M, Garcia S, Mancini J, Jammes Y, Courageot J, Lavieille JP, Feron F. Vitamin D3 potentiates myelination and recovery after facial nerve injury. Eur Arch Otorhinolaryngol. 2015 Oct;272(10):2815-23. doi: 10.1007/s00405-014-3305-y. Epub 2014 Sep 27. PMID 25261104
- [Background] Pomares G, Dap F, Dautel G. Complete section of proper palmar digital pedicles: Correlation between arterial patency and sensory recovery. Hand Surg Rehabil. 2017 Apr;36(2):136-140. doi: 10.1016/j.hansur.2016.12.001. Epub 2017 Mar 9. PMID 28325428
- [Background] Przybelski R, Agrawal S, Krueger D, Engelke JA, Walbrun F, Binkley N. Rapid correction of low vitamin D status in nursing home residents. Osteoporos Int. 2008 Nov;19(11):1621-8. doi: 10.1007/s00198-008-0619-x. Epub 2008 Apr 18. PMID 18421544
- [Background] Romagnoli E, Mascia ML, Cipriani C, Fassino V, Mazzei F, D'Erasmo E, Carnevale V, Scillitani A, Minisola S. Short and long-term variations in serum calciotropic hormones after a single very large dose of ergocalciferol (vitamin D2) or cholecalciferol (vitamin D3) in the elderly. J Clin Endocrinol Metab. 2008 Aug;93(8):3015-20. doi: 10.1210/jc.2008-0350. Epub 2008 May 20. PMID 18492750
- [Background] Shimokata H, Kuzuya F. Two-point discrimination test of the skin as an index of sensory aging. Gerontology. 1995;41(5):267-72. doi: 10.1159/000213693. PMID 8537010
- [Background] Shooter D. Use of two-point discrimination as a nerve repair assessment tool: preliminary report. ANZ J Surg. 2005 Oct;75(10):866-8. doi: 10.1111/j.1445-2197.2005.03557.x. PMID 16176227
- [Background] Taylor PN, Davies JS. A review of the growing risk of vitamin D toxicity from inappropriate practice. Br J Clin Pharmacol. 2018 Jun;84(6):1121-1127. doi: 10.1111/bcp.13573. Epub 2018 Apr 16. PMID 29498758
- [Background] Vieth R. Vitamin D supplementation, 25-hydroxyvitamin D concentrations, and safety. Am J Clin Nutr. 1999 May;69(5):842-56. doi: 10.1093/ajcn/69.5.842. PMID 10232622
- [Background] Vieth R. Why the optimal requirement for Vitamin D3 is probably much higher than what is officially recommended for adults. J Steroid Biochem Mol Biol. 2004 May;89-90(1-5):575-9. doi: 10.1016/j.jsbmb.2004.03.038. PMID 15225842
- [Background] Vieth R, Chan PC, MacFarlane GD. Efficacy and safety of vitamin D3 intake exceeding the lowest observed adverse effect level. Am J Clin Nutr. 2001 Feb;73(2):288-94. doi: 10.1093/ajcn/73.2.288. PMID 11157326
- [Background] Vieth R, Pinto TR, Reen BS, Wong MM. Vitamin D poisoning by table sugar. Lancet. 2002 Feb 23;359(9307):672. doi: 10.1016/S0140-6736(02)07814-5. No abstract available. PMID 11879864